CLINICAL TRIAL: NCT07040566
Title: Investigating Efficacious E-Cigarette Interventions and Cessation Effects on Cancer-Related Biomarkers: A Randomized Trial of Varenicline in Adults
Brief Title: A Trial of Varenicline for E-cigarette Cessation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000038513; 1R01CA296186-01 (NIH)
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: E-cigarette Use; Vaping; Nicotine Dependence
MeSH Terms: conditions — Vaping; Tobacco Use Disorder | interventions — Varenicline; BID protein, human

STUDY DESIGN:
Intervention Model Description: Adults who report regular e-cigarette use
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Varenicline (Experimental): Participants will randomly be assigned to 12-weeks of varenicline (titrated to 2mg daily) plus brief cessation advice with a counselor and self-management resources.
  Interventions: Drug: Varenicline 1mg BID
- Placebo (Placebo Comparator): Participants will randomly be assigned to 12-weeks of matching placebo plus brief cessation advice with a counselor and self-management resources.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline 1mg BID — 12 weeks following the standard titration of 1 mg, twice daily
  Arms: Varenicline
Drug: Placebo — Matching placebo twice daily
  Arms: Placebo

SUMMARY:
This is randomized, placebo-controlled clinical trial in treatment-seeking adults who report regular e-cigarette use to test the hypothesis that varenicline is efficacious for quitting e-cigarettes.

DETAILED DESCRIPTION:
Participants will randomly be assigned to 12-weeks of varenicline (titrated to 2mg daily) or matching placebo plus brief cessation advice from a counselor and self-management resources. All participants will also complete research assessments every 3 weeks during treatment and a final follow-up visit at week 26.

The primary objective is to test the efficacy of varenicline vs. placebo on e-cigarette quit rates. We will also evaluate predictors and moderators of outcomes and explore changes in health biomarkers following e-cigarette cessation treatment.

ELIGIBILITY:
Inclusion Criteria:

* report daily use of an e-cigarette containing nicotine
* live in Connecticut or South Carolina

Exclusion Criteria:

* regular use of other tobacco products besides e-cigarettes
* medical contraindications for varenicline use
* current treatment for tobacco cessation
* lack proficiency in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2030-07-30 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Abstinent From E-cigarette Use at Week 12 | Week 12
  7-day point-prevalence e-cigarette abstinence (PPA) at Week 12 defined as no ecigarette use [and no use of any combusted tobacco product], not even a puff, biochemically verified by saliva cotinine

SECONDARY OUTCOMES:
Number of Participants Abstinent From E-cigarette Use at Week 26 | Week 26
  7-day point-prevalence e-cigarette abstinence (PPA) at Week 26 defined as no ecigarette use [and no use of any combusted tobacco product], not even a puff, biochemically verified by saliva cotinine

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Fucito, PhD, Principal Investigator — Yale University; Benjamin Toll, PhD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Yale Cancer Center/Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Hollings Cancer Center at MUSC (HCC), Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared to an NIH data repository - the NIMH Data Archive
Supporting Information: Study Protocol, SAP
Access Criteria: Access to the data is managed by the NIMH Data Archive